CLINICAL TRIAL: NCT00071955
Title: A Phase II Study to Evaluate Safety and Efficacy of Specific Immunotherapy, Recombinant Idiotype Conjugated to KLH and GM-CSF Following the Anti-CD20 Antibody, Rituximab, in Previously Treated Patients With Follicular Non-Hodgkin's Lymphoma
Brief Title: Vaccine Therapy and Sargramostim After Rituximab in Treating Patients With Refractory or Progressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genitope Corporation (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269810; GENITOPE-2002-09; IUMC-0212-20
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2006-01

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — sargramostim

INTERVENTIONS:
Biological: autologous immunoglobulin idiotype-KLH conjugate vaccine
Biological: sargramostim

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Vaccines made from a person's cancer cells may make the body build an immune response to kill cancer cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood.

PURPOSE: Phase II trial to study the effectiveness of rituximab followed by vaccine therapy and sargramostim in treating patients who have refractory or progressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine progression-free survival in patients with refractory or progressive follicular non-Hodgkin's lymphoma treated with immediate or delayed autologous immunoglobulin idiotype-KLH conjugate vaccine and sargramostim after rituximab (groups I and II).
* Determine the immune response rate in patients treated with these regimens (groups I, II, and III).
* Determine the safety and toxicity of these regimens in these patients (groups I, II, and III).

OUTLINE: This is an open-label, multicenter study for patients previously registered on and confirmed ineligible for randomization in protocol Genitope-G2000-03.

Patients receive rituximab IV weekly for 4 weeks.

* Group I: The first 30 patients to achieve and maintain a partial response (PR) or better receive autologous immunoglobulin idiotype-KLH conjugate vaccine subcutaneously (SC) on day 1 and sargramostim SC on days 1-4 beginning 26 weeks after the last dose of rituximab. Treatment repeats every 2 weeks for 14 weeks (8 immunizations).
* Group II: All subsequent patients who achieve a PR or better receive autologous immunoglobulin idiotype-KLH conjugate vaccine and sargramostim SC as in group I beginning 13 weeks after the last dose of rituximab.
* Group III: Patients who are not eligible for group I or II and, in the investigator's opinion, are suitable candidates for immunization with autologous immunoglobulin idiotype-KLH conjugate vaccine and sargramostim SC receive the same treatment as groups I and II, beginning no more than 1 year after the last (fourth) dose of rituximab.

In all groups, treatment continues in the absence of unacceptable toxicity or emergence of an illness that may interfere with study assessments.

Patients are followed for initial response 8 weeks after completion of immunizations and then every 12 weeks for an additional year. Thereafter, all immunized patients will be followed every 6 months until receipt of first subsequent anti-lymphoma therapy.

PROJECTED ACCRUAL: Up to 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular center cell non-Hodgkin's lymphoma
* Stage III or IV disease at time of entry on Genitope-G2000-03
* At least 1 bidimensionally measurable lesion (1.5 cm X 1.5 cm) by radiography
* Previously registered on and confirmed to be ineligible for randomization on Genitope-G2000-03 by failing to achieve or maintain a complete or partial response after chemotherapy by CT scans of the chest, abdomen, and pelvis (and neck if there was palpable disease)
* Completed all 8 courses of chemotherapy (cyclophosphamide, vincristine, and prednisone [CVP]) per Genitope-G2000-03
* No intervening therapy for lymphoma (i.e., antibody, corticosteroids, or cytotoxic) between CVP and study entry
* No evidence of transformation (e.g., rapid tumor growth or increasing lactic dehydrogenase)
* No CNS involvement

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after the last immunization series
* HIV negative
* No history of autoimmune disease or conditions requiring treatment with immunosuppressive agents, including corticosteroids
* No other malignancy within the past 2 years except non-basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics
* At least 6 months since prior corticosteroids, including topical administration for any concurrent disease
* No concurrent chronic (more than twice monthly) corticosteroids (including topical or inhaled)

  * Transient use (prior to CT scan) or optical solutions allowed

Radiotherapy

* Prior radiotherapy to no more than 2 sites more than 13 weeks before rituximab is allowed

Surgery

* Not specified

Other

* No concurrent participation in other therapeutic clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03; Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in groups I and II and median PFS by Kaplan-Meier curves quarterly for 1 year and then twice a year after study completion

SECONDARY OUTCOMES:
Immune response rates in patients who received at least 4 immunizations by anti-idiotype antibody and anti-KLH antibody assays during every other immunization, last immunization, 2 and 8 weeks post immunization, and then quarterly for 1 year
Clinical response in patients who received at least 1 immunization in groups I and II by modified Cheson criteria post-immunization and then every 6 months for 1 year
Safety at the start of immunization, every 8 weeks during immunization, 2 and 8 weeks post immunization, and then quarterly for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Martha Mayo, PharmD, Study Chair — Genitope Corporation
Locations (11):
- United States (9):
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
- Canada (2):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Result] Timmerman JM, Vose JM, Czerwinski DK, Weng WK, Ingolia D, Mayo M, Denney DW, Levy R. Tumor-specific recombinant idiotype immunisation after chemotherapy as initial treatment for follicular non-Hodgkin lymphoma. Leuk Lymphoma. 2009 Jan;50(1):37-46. doi: 10.1080/10428190802563355. PMID 19125383